CLINICAL TRIAL: NCT03348046
Title: Post-Authorization Safety Study of Remsima® (Infliximab) in Rheumatoid Arthritis Patients in Jordan
Brief Title: Safety Study of Remsima® (Infliximab) in Rheumatoid Arthritis Patients in Jordan
Acronym: PASSRRA
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Other Study IDs: RMS-JOR-2015-01
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Infliximab; Remsima; Biosimilar; Autoimmune Disease; Rheumatoid Arthritis; Cohort Study; Disease modifying anti-rheumatic drugs; Tumor necrosis factor-alpha inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases | interventions — CT-P13

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Biosimilar Infliximab — A vial containing powder for concentrate for solution for infusion. Each vial contains: Infliximab 100 mg
  Other Names: Remsima®

SUMMARY:
The purpose of this observational study is to assess the safety and effectiveness of biosimilar Infliximab in patients with rheumatoid arthritis(RA) in Jordan where no visits or intervention(s) additional to the daily practice will be performed

DETAILED DESCRIPTION:
A multi-center, observational, prospective, cohort study to assess the safety and effectiveness of biosimilar Infliximab (Remsima®) in patients with rheumatoid arthritis in Jordan. Biologic naïve patients will receive Remsima® in accordance with standard medical care and the approved label and will be followed over a period of 34 weeks (8.5 months). Outcomes including occurrence of adverse events (AEs), mean changes in disease activity and health assessment in each cohort will be measured and compared

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Biologic naïve patients with active RA diagnosed according to the revised 1987 American College of Rheumatology (ACR) (Arnett et al. 1988) or 2010 ACR / European League Against Rheumatism (EULAR) Rheumatoid Arthritis classification criteria (Aletaha et al. 2010)
* Patients should be receiving a stable dose Methotrexate (MTX) for at least 3 months prior to enrolment, and still have active disease defined as erythrocyte sedimentation rate (ESR) ≥28 mm/h and swollen and tender joints ≥ 6
* Absence of tuberculosis demonstrated by negative chest X-ray

Exclusion Criteria:

* Patient <18 years
* Previous treatment with biologics
* Patients who meet any of the contraindications to the administration of infliximab
* Previous or concurrent malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from rheumatology outpatient clinics of 2 hospitals in Jordan
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) to Remsima® | 8.5 months
  Rate of AEs leading to permanent treatment discontinuation and rate of clinically relevant changes in laboratory tests will be calculated

SECONDARY OUTCOMES:
Mean changes in disease activity scores (DAS28)- Number of swollen joints | 8.5 months, changes between baseline and last visit will be compared between visits using repeated measure analyses
  The Disease Activity Score (DAS) measures the disease activity in patients with Rheumatoid Arthritis (RA). DAS28 is a validated simplified tool in which twenty-eight joints are measured. The number of swollen joints will be assessed.
Mean changes in disease activity scores (DAS28)-Number of tender joints | 8.5 months, changes between baseline and last visit will be compared between visits using repeated measure analyses
  The Disease Activity Score (DAS) measures the disease activity in patients with Rheumatoid Arthritis (RA). DAS28 is a validated simplified tool in which twenty-eight joints are measured. The number of tender joints will be assessed.
Mean changes in disease activity scores (DAS28)-ESR (Erythrocyte Sedimentation Rate) | 8.5 months, changes between baseline and last visit will be compared between visits using repeated measure analyses
  The Disease Activity Score (DAS) measures the disease activity in patients with Rheumatoid Arthritis (RA). DAS28 is a validated simplified tool in which twenty-eight joints are measured.
  ESR (Erythrocyte Sedimentation Rate) will be measured in mm/hr.
Mean changes in disease activity scores (DAS28)- Global assessment of disease activity on a 100 mm Visual Analogue Scale (VAS) | 8.5 months, changes between baseline and last visit will be compared between visits using repeated measure analyses
  The Disease Activity Score (DAS) measures the disease activity in patients with Rheumatoid Arthritis (RA). DAS28 is a validated simplified tool in which twenty-eight joints are measured.
  Patients will be asked to make a global assessment of disease activity on a 100 mm Visual Analogue Scale (VAS) measured by units on scale.
  Number of swollen and tender joints, Erythrocyte Sedimentation Rate and global assessment of disease activity on a 100 mm Visual Analogue Scale (VAS) are then fed into a complex mathematical formula to produce the overall disease activity score.
  The DAS28 provides a number on a scale from 0 to 10 indicating the current activity of the RA of the patient. A DAS28 above 5.1 means high disease activity whereas a DAS28 below 3.2 indicates low disease activity. Remission is achieved by a DAS28 lower than 2.6.
Mean changes in Disability Index of the Health Assessment Questionnaire (HAQ-DI) | 8.5 months, changes between baseline and last visit will be compared between visits using repeated measure analyses
  The Health assessment questionnaire disability index (HAQ-DI) is a questionnaire for the assessment of Rheumatoid Arthritis. The reported data from patients include the amount of difficulty they have in performing some of their activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3).

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Prince Hamza Hospital, Amman
  - Jordan University of Science and Technology- King Abdallah University Hospital, Irbid

IPD SHARING:
Plan to Share IPD: No